CLINICAL TRIAL: NCT01247779
Title: Assessment of Perioperative Morbidity in Gyneco-oncology According to the Surgical Approach : Coelioscopy Versus Robot-assisted Coelioscopy
Brief Title: Perioperative Morbidity in Gyneco-oncology According to the Procedure : Coelioscopy Versus Robot-assisted Coelioscopy
Acronym: ROBO-GYN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Oscar Lambret (Other)
Collaborators: CRG : Groupe Francophone de Chirurgie Robotique en Gynécologie (Unknown); National Cancer Institute, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ROBOGYN - 1004; 2010-A00605-34 (Other: IDRCB Number (ANSM_DEDIM))
Record Dates: First submitted 2010-11-19; First posted 2010-11-24 (Estimated); Last update posted 2019-03-08 (Actual); Status verified 2019-03

CONDITIONS: Cervical Cancer; Uterus Cancer; Ovarian Cancer
Keywords: gynecology; oncology; coelioscopy; robot; morbidity
MeSH Terms: conditions — Uterine Cervical Neoplasms; Uterine Neoplasms; Ovarian Neoplasms; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Coelioscopy (Active Comparator): gynecologic surgery - standard coelioscopy
  Interventions: Procedure: gynecologic surgery - standard coelioscopy
- Robot-assisted coelioscopy (Experimental): gynecologic surgery - robot assisted coelioscopy
  Interventions: Procedure: gynecologic surgery - robot assisted coelioscopy

INTERVENTIONS:
Procedure: gynecologic surgery - standard coelioscopy — lymphadenectomy; hysterectomy; nerve sparing; enlarged trachelectomy; omentectomy; appendicectomy; pelvectomy
  Arms: Standard Coelioscopy
Procedure: gynecologic surgery - robot assisted coelioscopy — lymphadenectomy; hysterectomy; nerve sparing; enlarged trachelectomy; omentectomy; appendicectomy; pelvectomy
  Arms: Robot-assisted coelioscopy

SUMMARY:
The purpose of this study is to compare perioperative morbidity of coelioscopy versus robot-assisted coelioscopy in cervical cancer, uterus cancer and ovarian cancer.

DETAILED DESCRIPTION:
Laparoscopic surgery, also called minimally invasive surgery (MIS), is a surgical method less invasive than classical laparoscopic open procedure. Particularly, MIS is used for resection of some gynecological cancer such as endometrial cancer, cervical cancer or ovarian cancer. Several studies demonstrated that MIS induce less surgical complications (bleeding, infections, post-operative pains...), shorter hospitalization time, earlier recovery of activity and better quality of life than laparoscopic open procedure.

However, MIS is the selected method in only 9 to 25 % of gynecologic cancer surgery in France. This is likely due to the longer learning curve of MIS compared to laparoscopic open procedure.

In 2001 the FDA allowed the use of robot assisted laparoscopic surgery (RALS). This technique adds some advantage to laparoscopic surgery. Indeed, surgeon operates with better precision while seated comfortably at a computer console viewing a 3-D image of the surgical field. Moreover learning curve of RALS is shorter than MIS. Comparative studies between RALS and MIS demonstrate an equivalence of these techniques for operation length and bleeding. However for surgery linked complications and time for recovery of activity, RALS had better results than MIS.

Despite its expensive cost, RALS is now commonly used in North America (90% of prostatectomy and 40% of cancer linked hysterectomy). However RALS need to be evaluated in a randomized clinical trial before it's acceptation in gyneco-oncology in France.

Thus, the purpose of the ROBOGYN clinical trial is to compare clinical benefit of RALS and MIS in a randomized study for patients with cancer of cervix, uterus or ovary.

ELIGIBILITY:
Inclusion Criteria:

* patient with uterus cancer depending on hysterectomy ± pelvic lymphadenectomy or a restadification
* patient with cervical cancer depending on enlarged colpo-hysterectomy ± pelvic lymphadenectomy or a surgery after concomitant radiochemotherapy, or lombo aortic lymphadenectomy for a locally advanced cancer, or a restadification
* patient with cervical cancer depending on a restadification
* patient aged over 18 years
* previous antitumor treatment allowed but necessarily disrupted 20 days before inclusion
* WHO score equal or inferior to 3
* cirrhosis-related Child-Pugh score under or equal to A7 are allowed
* life expectancy equal or superior to 12 weeks
* patient affiliated to health insurance
* dated and signed informed consent

Exclusion Criteria:

* metastatic disease
* pregnant or breastfeeding woman
* patient unable to proceed follow-up visit, because of geographic, social or mental reasons

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 386 (Actual)
Dates: Start 2010-12 (Actual); Primary Completion 2016-03 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Perioperative morbidity at six months | six months after surgery
  To estimate the rate of complications within the first six months after surgery, according to the Clavien-Dindo and NCI CTCAE-v4.0 grading scales

SECONDARY OUTCOMES:
Anesthesic and ventilator parameters | every 30 min during the surgery
  Description of anesthesic and ventilator parameters
Post-operative analgesia | at 24h, 48h after sugery and until discharge
  collect of antalgic treatments
Surgeon's ergonomy | every hour during surgery (Borg scale), and at the end of intervention (NASA-TLX scale)
  according to Borg and NASA-TLX scales
Patient-reported survey of patient health | until 2 years after surgery
  36-item short form health Survey (SF36) : Scoring is a two-step process. First, numeric values of all items are recoded per the scoring key (for example, values are 0/100, or 0/25/50/75/100 depending the items). All items are scored so that a high score defines a more favorable health state. Each item is scored on a 0 to 100 range so that the lowest and highest possible scores are 0 and 100, respectively. Scores represent the percentage of total possible score achieved. In step 2, items in the same scale are averaged together to create the 8 scale scores: physical functioning, Role functioning/physical, Role functioning/emotional, Energy/fatigue, Emotional well-being, Social functioning, Pain, General health, Health change. Scale scores represent the average for all items in the scale that the respondent answered.
Description of surgical procedures | during surgery
  operative time (overall intervention, incision or "skin-to-skin", robot).
Progression-free survival | until 2 years after surgery
  delay between the date of randomization and the date of the following event: local relapse, regional relapse, metastasis or death.
Anatomopathology | during surgery
  rate of exeresis with histologically healthy resection margins (R0), number of lymph nodes removed.

CONTACTS AND LOCATIONS:
Overall Officials: Fabrice NARDUCCI, MD, Principal Investigator — Centre Oscar Lambret, Lille; Eric LAMBAUDIE, MD, Study Director — Institut Paoli-Calmettes
Locations (17):
- France (17):
  - CHU Bordeaux, Hôpital Saint-André, Bordeaux
  - Polyclinique Bordeaux Nord Aquitaine, Bordeaux
  - Centre Oscar Lambret, Lille
  - CHRU Lille, Hôpital Jeanne de Flandres, Lille
  - CHU Limoges, Limoges
  - Institut Paoli Calmette, Marseille
  - CHU Nîmes, Nîmes
  - Polyclinique KenVal, Nîmes
  - Hôpital Européen Georges Pompidou, Paris
  - Polyclinique Courlancy, Reims
  - Centre hospitalier de Roubaix, Roubaix
  - Institut de Cancérologie de l'Ouest Site René Gauducheau, Saint-Herblain
  - Institut Claudius Regaud, Toulouse
  - CHU Rangueil, Toulouse
  - CHRU de Tours, Tours
  - Centre Hospitalier de Valenciennes, Valenciennes
  - Centre Alexis Vautrin, Vandœuvre-lès-Nancy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Narducci F, Bogart E, Hebert T, Gauthier T, Collinet P, Classe JM, Lecuru F, Delest A, Motton S, Conri V, Ferrer C, Marchal F, Ferron G, Probst A, Thery J, Le Deley MC, Lefebvre D, Francon D, Leblanc E, Lambaudie E. Severe perioperative morbidity after robot-assisted versus conventional laparoscopy in gynecologic oncology: Results of the randomized ROBOGYN-1004 trial. Gynecol Oncol. 2020 Aug;158(2):382-389. doi: 10.1016/j.ygyno.2020.05.010. Epub 2020 May 25. PMID 32467054